CLINICAL TRIAL: NCT03935984
Title: Improving the Sensitivity of Sestamibi SPECT-CT Parathyroid Scan with Calcitonin Pre-treatment for Primary Hyperparathyroidism
Brief Title: Calcitonin Pre-treatment to Improve SPECT-CT Sensitivity
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Joseph Sferra (Other)
Collaborators: University of Toledo Health Science Campus (Other)
Responsible Party: Sponsor-Investigator, Joseph Sferra, Chief of Surgery, ProMedica Health System
Organization: ProMedica Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-018
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Primary Hyperparathyroidism; Hypercalcemia
MeSH Terms: conditions — Hyperparathyroidism, Primary; Hypercalcemia | interventions — Calcitonin; salmon calcitonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): All subjects in this arm will be treated with calcitonin 200IU 2x per day for 2 days, then 1x on day of SPECT-CT imaging
  Interventions: Drug: Calcitonin

INTERVENTIONS:
Drug: Calcitonin — Treatment with calcitonin to lower high calcium levels prior to reimaging exam
  Other Names: Miacalcin

SUMMARY:
Patients with biochemically confirmed primary hyperparathyroidism and non-localizing SPECT-CT exam within the past year will be included. Subjects will be treated with calcitonin to lower calcium levels immediately prior to reimaging. The goal of this study is to determine whether lowering calcium will improve uptake/retention of sestamibi and improve sensitivity of SPECT-CT to localize parathyroid adenoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary hyperparathyroidism
* Non-localizing SPECT-CT performed within 365 days prior to consent to participate in study
* Patient desires surgical intervention for treatment of PHPT
* No contraindications to 99mTC-Sestamibi
* No contraindications to treatment with calcitonin
* Serum calcium level prior to non-localizing SPECT-CT is ≥10.5 mg/dL
* Patient consents to participate and undergo second SPECT-CT for purposes of research

Exclusion Criteria:

* Previous surgery to the neck, including resection of parathyroid tissue, except where end organ damage is present and further surgical intervention is medically necessary
* Contraindication to 99mTC-Sestamibi SPECT-CT as evidenced by allergic reaction or adverse event during index SPECT-CT
* Allergy to calcitonin
* Hypocalcemia (contraindication to calcitonin)
* Vitamin D deficiency (contraindication to calcitonin)
* Previous treatment with radioactive iodine
* New prescription of thyroid medication (levothyroxine, armour thyroid tablets, etc. must be taken at time of index scan and research scan)
* Lithium exposure within one year of SPECT-CT (index and research scans)
* Secondary hyperparathyroidism
* Benign familial hypocalciuric hypercalcemia
* Known malignancy, particularly multiple endocrine neoplasia
* New prescription of thiazide diuretic, (thiazide diuretic must have been taken at the time of index scan and second scan)
* Currently taking calcium channel blockers
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2019-05-29 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of SPECT-CT | one year
  conversion rate from non-localizing to localizing exam

SECONDARY OUTCOMES:
Surgical Approach | 6 months
  Rate of minimally-invasive surgery compared to four gland exploration
Success Rate | 6 months from surgery
  Rate of patients in whom surgical intervention was successful in curing hyperparathyroidism

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Sferra, MD, Principal Investigator — University of Toledo College of Medicine
Locations (1):
- ProMedica Toledo Hospital, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No